CLINICAL TRIAL: NCT01759589
Title: Sevoflurane Alone and Propofol With or Without Remifentanil in Electroconvulsive Therapy
Brief Title: Three Anaesthesic Method in Electroconvulsive Theraphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zekine Begec, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Inonu University Anesthesia; Inonu University (Other: Inonu University)
Record Dates: First submitted 2012-12-14; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Anesthesia
Keywords: electroconvulsive therapy,sevoflurane,propofol,remifentanil
MeSH Terms: interventions — Propofol; Remifentanil; Analgesics, Opioid; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- propofol (Group P) (Placebo Comparator): The patients in Group P received 1 mg/kg propofol IV (over 15 sec) during anesthesia induction
  Interventions: Drug: Propofol
- remifentanil and propofol (Group R) (Active Comparator): Patients in Group R received remifentanil 1 µg/kg IV (over 60 sec) and 0.5 mg/kg propofol IV (over 15 sec)during anesthesia induction
  Interventions: Drug: Remifentanil and propofol
- sevoflurane (Group S) (Active Comparator): In Group S, sevoflurane was started at 6% for induction and continued at 1% until the electrical stimulus was delivered, at which time it was stopped.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — 1 mg/kg propofol IV (over 15 sec) during anesthesia induction
  Other Names: Intravenous anesthetic agent
  Arms: propofol (Group P)
Drug: Remifentanil and propofol — 1 µg/kg IV (over 60 sec)remifentanil and 0.5 mg/kg propofol IV (over 15 sec)during anesthesia induction
  Other Names: Opioid and intravenous anesthetic agent
  Arms: remifentanil and propofol (Group R)
Drug: Sevoflurane — Sevoflurane was started at 6% for induction and continued at 1% until the electrical stimulus was delivered
  Other Names: Volatil anesthetic
  Arms: sevoflurane (Group S)

SUMMARY:
To compare the effectiveness of three different anesthetic regimens (propofol, remifentanil-propofol and sevoflurane in ECT.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of three different anesthetic regimens (propofol, remifentanil-propofol and sevoflurane) with respect to seizure duration, postictal suppression index, early and midictal amplitude, hemodynamic variables and recovery profiles in ECT.

ELIGIBILITY:
Inclusion Criteria:

* Upremedicated ASA I-II (American Society of Anesthesiologists's physical status) patients,
* Patients scheduled for six ECT sessions for a variety of psychiatric conditions (major depression, schizophrenia)

Exclusion Criteria:

* Involuntary patient status
* Patients with known or self-declared needle or mask phobia
* Pregnancy
* Asthma
* Cerebrovascular disease,
* History of myocardial infarction in the previous 6 months,
* Atrial fibrillation or flutter,heart block,
* A known or family history of reactions to the study drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Seizure duration | The patients were observed about seizure up to ten minutes after electrical stimulation
  After anesthesia induction patients were administered electrical stimulation and seizure duration were measured.

SECONDARY OUTCOMES:
postictal suppression index | completing seizure in one hour
  After anesthesia induction, patients were administered electrical stimulation. Then, postictal suppression index, a parameter that shows seizure quality, was determined from seizure records.
Recovery parameters (spontaneous breathing, eye opening, and obeying of verbal commands) | after seizure in one hour in operation room.
  The time from the end of succinylcholine administration to the recovery of spontaneous breathing, eye opening, and obeying of verbal commands were recorded.
Hemodynamic variables | Before administration of the study medications (t0), and at 1 (t1), 3 (t2), and 10 (t3) minutes after the seizure ended.
  During perioperative period:
  Before administration of the study medications (t0), and at 1 (t1), 3 (t2), and 10 (t3) minutes after the seizure ended.

CONTACTS AND LOCATIONS:
Overall Officials: Zekine Begec, Study Director
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Toprak HI, Gedik E, Begec Z, Ozturk E, Kaya B, Ersoy MO. Sevoflurane as an alternative anaesthetic for electroconvulsive therapy. J ECT. 2005 Jun;21(2):108-10. doi: 10.1097/01.yct.0000166633.73555.28. PMID 15905753